## AGE AND SEX DIFFERENCES IN THE METABOLIC RESPONSE TO EXERCISE

Date: 24th March 2023



## CONSENT FORM FOR ADULT PARTICIPANTS IN RESEARCH STUDIES

Please complete this form after you have read the Information Sheet and/or listened to an explanation about the research.

Title of Study: Age and sex differences in the metabolic response to exercise

**Department:** UCL Great Ormond Street Institute of Child Health

Name and Contact Details of the Researcher(s): Evelyn Maniaki (<a href="Evelyn.Maniaki.20@ucl.ac.uk">Evelyn.Maniaki.20@ucl.ac.uk</a>), Andy Galbraith (A.J.Galbraith@uel.ac.uk), and Jonathan Wells (Jonathan.Wells@ucl.ac.uk)

Name and Contact Details of the Principal Researcher: Jonathan Wells (<u>Jonathan.Wells@ucl.ac.uk</u>)

Name and Contact Details of the UCL Data Protection Officer: Alexandra Potts (data-protection@ucl.ac.uk)

This study has been approved by the UCL Research Ethics Committee (Project ID number 0326/020) and the UEL Research Ethics Committee (Project ID number 2223-0081).

Thank you for considering taking part in this research. The person organising the research must explain the project to you before you agree to take part. If you have any questions arising from the Information Sheet or explanation already given to you, please ask the researcher before you decide whether to join in. You will be given a copy of this Consent Form to keep and refer to at any time.

For your reference, the exclusion criteria are as follows:

- 1. Having a chronic illness.
- 2. Having a disease, disability or other condition that would impair participation in physical activity.
- 3. Having an implanted cardiac pacemaker, defibrillator, or other electronic medical devices.
- 4. Taking prescription medication one or more days every week over the past 3 months.
- 5. Related by blood to another participant.
- 6. Not willing at the time of recruitment to undergo blood sampling.
- 7. Pregnancy/breastfeeding.
- 8. Being a professional athlete.
- 9. Not being physically active.
- 10. Being a shift worker (night shift work for three or more days per week on more than two occasions in the six months before the visit day).
- 11. Recent weight loss of more than 5% of weight in the last 6 months.
- 12. Having a body mass index outside the range of 19 to 24.5.
- 13. Smoking/vaping.
- 14. Alcohol intake above an NHS questionnaire cut-off.
- 15. Regular use of recreational drugs.
- 16. Exhibiting any symptoms related to COVID-19 during a period.
- 17. Not having reached menopause (i.e., your period has not stopped for 12 months or more for women aged 53-57 only).

I confirm that I understand that by ticking/initialling each box below I am consenting to this element of the study. I understand that it will be assumed that unticked/initialled boxes means that I DO NOT consent to that part of the study. I understand that by not giving consent for any one element that I may be deemed ineligible for the study.

| | | Tick |
|---|---|---|
| | | Box |
| | I confirm that I have read and understood the Information Sheet for the above study. I have had | |
| 1. | an opportunity to consider the information and what will be expected of me, and I have also had | |
| | the opportunity to ask questions which have been answered to my satisfaction. | |
| 2. | I confirm that I will have my saliva collected on three occasions. | |
| 3. | I confirm that I will have blood samples collected on three occasions via venepuncture. | |
| 4. | I confirm that I will have my weight, height, waist, and hip circumference measured. | |
| 5. | I confirm that I will have my body composition measured. | |
| 6. | I confirm that I will drink deuterium-labelled water. | |
| 7. | I confirm that I will have my heart rate measured. | |
| 8. | I confirm that I will have my blood pressure measured. | |
| 9. | I confirm that I will undertake a treadmill exercise challenge. | |
| 10. | I confirm that I will have my expired breath measured. | |
| 44 | I confirm that I will complete two questionnaires assessing my mood, appetite, feeling of | |
| 11. | tiredness as well as verbal learning on three occasions. | |
| 12. | I understand that I will be able to withdraw my data up to 4 weeks after the visit. | |
| | I consent to participate in the study. I understand that my personal information (first and last | |
| | name, full postal address, email address, phone number, date of birth, sex, ethnic origin, and | |
| 13. | health) will be used for the purposes explained to me. I understand that according to data | |
| | protection legislation, 'public task' will be the lawful basis for processing my <i>personal</i> data and | |
| | 'scientific and historical research or statistical purposes' for special category personal data. | |
| | Use of the information for this project only | |
| | • I understand that all personal information will remain confidential and that all efforts will be | |
| | made to ensure I cannot be identified. | |
| | • I understand that my data gathered in this study will be stored anonymously and securely. It | |
| 14. | | |
| | • I understand that confidentiality will be respected unless there are compelling and legitimate | |
| | reasons for this to be breached. If this was the case, we would inform you of any decision | |
| | that might limit your confidentiality. | |
| 15. | I understand that my information may be subject to review by responsible individuals from the | |
| 10. | University for monitoring and audit purposes. | |
| | I understand that my participation is voluntary and that I am free to withdraw at any time | |
| | without giving a reason, without my legal rights being affected. | |
| 16. | • I understand that if I decide to withdraw, any personal data I have provided up to that point | |
| | will be deleted unless I agree otherwise. | |
| | I understand the potential risks of participating and the support that will be available to me | |
| 17. | should I become distressed during the course of the research. | |
| 10 | | |
| 18. | I understand the direct/indirect benefits of participating. | |
| 19. | I understand that the data will not be made available to any commercial organisations but is | |
| | solely the responsibility of the researchers undertaking this study. | |
| 20. | I understand that I will not benefit financially from this study or from any possible outcome it may | |
| | result in in the future. | |
| 21. | I agree that my anonymised research data may be used by others for future research. No one will | |
| | be able to identify you when this data is shared. | |

| Thereby confirm that I understand the inclusion criteria as detailed in the Information Sheet and explained to me by the researcher. I hereby confirm that: (a) I understand the exclusion criteria as detailed in the Information Sheet and explained to me by the researcher (Having a chronic illness; Having a disease, disability or other condition that would impair participation in physical activity; Having an implanted cardiac pacemaker, defibrillator, or other electronic medical device; Taking prescription medication one or more days every week over the past 3 months; Related by blood to another participant; Not willing at the time of recruitment to undergo blood sampling; Pregnancy / breastfeeding; Being a professional athlete; Not being physically active; Being a shift worker (night shift work for three or more days per week on more than two occasions in the six months before the visit day); Recent weight loss of more than 5% of weight in the last 6 months; Having a body mass index outside the range of 19 to 24.5; Smoking vaping; Alcohol intake above NH5 questionnaire cut-off; Regular use of recreational drugs; Exhibiting any symptoms related to COVID-19 during a period; Not having reached menopause [i.e., your period has not stopped for 12 months or more — for women aged 53-57 only]) (b) I do not fall under the exclusion criteria. 25. I have informed the researcher of any other research in which I am currently involved or have been involved in during the past 12 months. 26. I am aware of who I should contact if I wish to lodge a complaint. 27. I voluntarily agree to take part in this study. 28. I would be happy for the data I provide to be archived at the UCL Research Data Repository. • I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. • I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Resea | 1 hereby confirm that I understand the inclusion criteria as detailed in the Information Sheet and explained to me by the researcher. 1 hereby confirm that: (a) I understand the exclusion criteria as detailed in the Information Sheet and explained to me by the researcher (Having a chronic illness; Having a disease, disability or other condition that would impair participation in physical activity; Having an implanted cardiac pacemaker, defibrillator, or other electronic medical device; Taking prescription medication one or more days every week over the past 3 months; Related by blood to another participant; Not willing at the time of recruitment to undergo blood sampling; Pregnancy / breastfeeding; Being a professional athlete; Not being physically active; Being a shift worker (night shift work for three or more days per week on more than two occasions in the six months before the visit day); Recent weight loss of more than 5% of weight in the last 6 months; Having a body mass index outside the range of 19 to 24.5; Smoking vaping; Alcohol intake above NHS questionnaire cut-off; Regular use of recreational drugs; Exhibiting any symptoms related to COVID-19 during a period; Not having reached menopause [i.e., your period has not stopped for 12 months or more – for women aged 53-57 only]) (b) I do not fall under the exclusion criteria. 1 have informed the researcher of any other research in which I am currently involved or have been involved in during the past 12 months. 25. | 1 | 22. | I understand that the information I have submitted may be published as a report and I wish to receive a copy of it. Yes/No | | |
|---|---|---|---|---|---|---|
| explained to me by the researcher. I hereby confirm that: (a) I understand the exclusion criteria as detailed in the Information Sheet and explained to me by the researcher (Having a chronic illness; Having a disease, disability or other condition that would impair participation in physical activity; Having an implanted cardiac pacemaker, defibrillator, or other electronic medical device; Taking prescription medication one or more days every week over the past 3 months; Related by blood to another participant; Not willing at the time of recruitment to undergo blood sampling; Pregnancy / breastfeeding; Being a professional athlete; Not being physically active; Being a shift worker (night shift work for three or more days per week on more than two occasions in the six months before the visit day); Recent weight loss of more than 5% of weight in the last 6 months; Having a body mass index outside the range of 19 to 24.5; Smoking vaping; Alcohol intake above NHS questionnaire cut-off; Regular use of recreational drugs; Exhibiting any symptoms related to COVID-19 during a period; Not having reached menopause [i.e., your period has not stopped for 12 months or more — for women aged 53-57 only]) (b) I do not fall under the exclusion criteria. 1 have informed the researcher of any other research in which I am currently involved or have been involved in during the past 12 months. 25. I am aware of who I should contact if I wish to lodge a complaint. 27. I voluntarily agree to take part in this study. Use of information for this project and beyond: • I would be happy for the data I provide to be archived at the UCL Research Data Repository. • I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. • I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These res | 23. explained to me by the researcher. Thereby confirm that: | Explained to me by the researcher. | | · | inclusion criteria as detailed in the Information Sheet and | |
| I hereby confirm that: (a) I understand the exclusion criteria as detailed in the Information Sheet and explained to me by the researcher (Having a chronic illness; Having a disease, disability or other condition that would impair participation in physical activity; Having an implanted cardiac pacemaker, defibrillator, or other electronic medical device; Taking prescription medication one or more days every week over the past 3 months; Related by blood to another participant; Not willing at the time of recruitment to undergo blood sampling; Pregnancy / breastfeeding; Being a professional athlete; Not being physically active; Being a shift worker (night shift work for three or more days per week on more than two occasions in the six months before the visit day); Recent weight loss of more than 5% of weight in the last 6 months; Having a body mass index outside the range of 19 to 24.5; Smoking vaping; Alcohol intake above NHS questionnaire cut-off; Regular use of recreational drugs; Exhibiting any symptoms related to COVID-19 during a period; Not having reached menopause [i.e., your period has not stopped for 12 months or more – for women aged 53-57 only]) (b) I do not fall under the exclusion criteria. Thave informed the researcher of any other research in which I am currently involved or have been involved in during the past 12 months. | I hereby confirm that: (a) I understand the exclusion criteria as detailed in the Information Sheet and explained to me by the researcher (Having a chronic illness; Having a disease, disability or other condition that would impair participation in physical activity; Having an implanted cardiac pacemaker, defibrillator, or other electronic medical device; Taking prescription medication one or more days every week over the past 3 months; Related by blood to another participant; Not willing at the time of recruitment to undergo blood sampling; Pregnancy / breastfeeding; Being a professional athlete; Not being physically active; Being a shift worker (night shift work for three or more days per week on more than two occasions in the six months before the visit day); Recent weight loss of more than 5% of weight in the last 6 months; Having a body mass index outside the range of 19 to 24.5; Smoking vaping; Alcohol intake above NHS questionnaire cut-off; Regular use of recreational drugs; Exhibiting any symptoms related to COVID-19 during a period; Not having reached menopause [i.e., your period has not stopped for 12 months or more — for women aged 53-57 only]) (b) I do not fall under the exclusion criteria. 1 have informed the researcher of any other research in which I am currently involved or have been involved in during the past 12 months. 25. I am aware of who I should contact if I wish to lodge a complaint. 27. I voluntarily agree to take part in this study. 28. I would be happy for the data I provide to be archived at the UCL Research Data Repository. 1 understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. 1 understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians. | I hereby confirm that: | 23. | | | |
| 25. I have informed the researcher of any other research in which I am currently involved or have been involved in during the past 12 months. 26. I am aware of who I should contact if I wish to lodge a complaint. 27. I voluntarily agree to take part in this study. Use of information for this project and beyond: I would be happy for the data I provide to be archived at the UCL Research Data Repository. I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians. | 25. I have informed the researcher of any other research in which I am currently involved or have been involved in during the past 12 months. 26. I am aware of who I should contact if I wish to lodge a complaint. 27. I voluntarily agree to take part in this study. Use of information for this project and beyond: I would be happy for the data I provide to be archived at the UCL Research Data Repository. I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians. | 25. I have informed the researcher of any other research in which I am currently involved or have been involved in during the past 12 months. 26. I am aware of who I should contact if I wish to lodge a complaint. 27. I voluntarily agree to take part in this study. Use of information for this project and beyond: I would be happy for the data I provide to be archived at the UCL Research Data Repository. I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians. Would like your contact details to be retained so that you can be contacted in the future by UCL research like to invite you to participate in follow up studies to this project, or in future studies of a similar nature exappropriate box below. Yes, I confirm that I am willing to be contacted in this way No, I do not confirm that I am willing to be contacted | | I hereby confirm that: (a) I understand the exclusion criteria by the researcher (Having a chroni would impair participation in physidefibrillator, or other electronic mays every week over the past 3 mat the time of recruitment to under professional athlete; Not being physically three or more days per week on may); Recent weight loss of more tindex outside the range of 19 to 24 questionnaire cut-off; Regular use COVID-19 during a period; Not have for 12 months or more — for women. | ic illness; Having a disease, disability or other condition the ical activity; Having an implanted cardiac pacemaker, edical device; Taking prescription medication one or more nonths; Related by blood to another participant; Not willing blood sampling; Pregnancy / breastfeeding; Being a sysically active; Being a shift worker (night shift work for more than two occasions in the six months before the visit han 5% of weight in the last 6 months; Having a body mas 4.5; Smoking vaping; Alcohol intake above NHS of recreational drugs; Exhibiting any symptoms related to ving reached menopause [i.e., your period has not stoppe en aged 53-57 only]) | e ng |
| been involved in during the past 12 months. 26. I am aware of who I should contact if I wish to lodge a complaint. 27. I voluntarily agree to take part in this study. Use of information for this project and beyond: I would be happy for the data I provide to be archived at the UCL Research Data Repository. I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians. | been involved in during the past 12 months. 26. I am aware of who I should contact if I wish to lodge a complaint. 27. I voluntarily agree to take part in this study. Use of information for this project and beyond: I would be happy for the data I provide to be archived at the UCL Research Data Repository. I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians. | been involved in during the past 12 months. 26. I am aware of who I should contact if I wish to lodge a complaint. 27. I voluntarily agree to take part in this study. Use of information for this project and beyond: I would be happy for the data I provide to be archived at the UCL Research Data Repository. I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians. Would like your contact details to be retained so that you can be contacted in the future by UCL research like to invite you to participate in follow up studies to this project, or in future studies of a similar nature appropriate box below. Yes, I confirm that I am willing to be contacted in this way No, I do not confirm that I am willing to be contacted | | ` ' | | |
| 26. I am aware of who I should contact if I wish to lodge a complaint. 27. I voluntarily agree to take part in this study. Use of information for this project and beyond: I would be happy for the data I provide to be archived at the UCL Research Data Repository. I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians. | 26. I am aware of who I should contact if I wish to lodge a complaint. 27. I voluntarily agree to take part in this study. Use of information for this project and beyond: I would be happy for the data I provide to be archived at the UCL Research Data Repository. I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians. | 26. I am aware of who I should contact if I wish to lodge a complaint. 27. I voluntarily agree to take part in this study. Use of information for this project and beyond: I would be happy for the data I provide to be archived at the UCL Research Data Repository. I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians. Would like your contact details to be retained so that you can be contacted in the future by UCL research in the invite you to participate in follow up studies to this project, or in future studies of a similar nature exappropriate box below. Yes, I confirm that I am willing to be contacted in this way No, I do not confirm that I am willing to be contacted | 25. | · | • | |
| 27. I voluntarily agree to take part in this study. Use of information for this project and beyond: I would be happy for the data I provide to be archived at the UCL Research Data Repository. I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians. | 27. I voluntarily agree to take part in this study. Use of information for this project and beyond: I would be happy for the data I provide to be archived at the UCL Research Data Repository. I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians. Vould like your contact details to be retained so that you can be contacted in the future by UCL researchers in the project, or in future studies of a similar nature. | 27. I voluntarily agree to take part in this study. Use of information for this project and beyond: I would be happy for the data I provide to be archived at the UCL Research Data Repository. I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians. I would like your contact details to be retained so that you can be contacted in the future by UCL researches appropriate box below. Yes, I confirm that I am willing to be contacted in this way No, I do not confirm that I am willing to be contacted | 26 | _ : | | $\vdash$ |
| Use of information for this project and beyond: I would be happy for the data I provide to be archived at the UCL Research Data Repository. I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians. | Use of information for this project and beyond: I would be happy for the data I provide to be archived at the UCL Research Data Repository. I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians. I would like your contact details to be retained so that you can be contacted in the future by UCL researchers in the fu | Use of information for this project and beyond: I would be happy for the data I provide to be archived at the UCL Research Data Repository. I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians. I would like your contact details to be retained so that you can be contacted in the future by UCL research like to invite you to participate in follow up studies to this project, or in future studies of a similar nature appropriate box below. Yes, I confirm that I am willing to be contacted in this way No, I do not confirm that I am willing to be contacted | | | | |
| <ul> <li>I would be happy for the data I provide to be archived at the UCL Research Data Repository.</li> <li>I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below.</li> <li>I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians.</li> </ul> | <ul> <li>I would be happy for the data I provide to be archived at the UCL Research Data Repository.</li> <li>I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below.</li> <li>I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians.</li> </ul> vould like your contact details to be retained so that you can be contacted in the future by UCL researchers in volume to participate in follow up studies to this project, or in future studies of a similar nature. | I would be happy for the data I provide to be archived at the UCL Research Data Repository. I understand that my personal contact details will not be retained once the data collection has finished, unless I agree to be contacted for potential future studies as outlined below. I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be graduate students or statisticians. vould like your contact details to be retained so that you can be contacted in the future by UCL research like to invite you to participate in follow up studies to this project, or in future studies of a similar nature appropriate box below. Yes, I confirm that I am willing to be contacted in this way No, I do not confirm that I am willing to be contacted | | , , | | |
| ke to invite you to participate in follow up studies to this project, or in future studies of a similar nature | like to invite you to participate in follow up studies to this project, or in future studies of a similar natu | like to invite you to participate in follow up studies to this project, or in future studies of a similar nature appropriate box below. Yes, I confirm that I am willing to be contacted in this way No, I do not confirm that I am willing to be contacted | 28. | <ul> <li>has finished, unless I agree to be contacted for potential future studies as outlined below.</li> <li>I understand that other authenticated researchers will have access to my anonymised data which will be available at the UCL Research Data Repository. These researchers may be</li> </ul> | | |
| appropriate box below. | | No, I do not confirm that I am willing to be contacted | 26.<br>27.<br>28.<br>would<br>like to | been involved in during the past 12 mo I am aware of who I should contact if I I voluntarily agree to take part in this st Use of information for this project and I would be happy for the data I pro I understand that my personal contact has finished, unless I agree to be contact which will be available at the UCL R graduate students or statisticians. Iike your contact details to be retained invite you to participate in follow up | wish to lodge a complaint. tudy. beyond: vide to be archived at the UCL Research Data Repository. tact details will not be retained once the data collection ontacted for potential future studies as outlined below. ted researchers will have access to my anonymised data Research Data Repository. These researchers may be | . researc |